CLINICAL TRIAL: NCT00803673
Title: A Single Centre, Randomized, Double-blind, Dose Ascending, Placebo-controlled Study, in Two Parts, to Evaluate the Safety, Tolerability and Pharmacokinetics of Escalating Single and Repeat Inhaled Doses of GSK573719 and Placebo Formulated With the Excipient Magnesium Stearate, in Healthy Subjects and in a Healthy Population of Cytochrome P450 Isoenzyme 2D6 Poor Metabolisers.
Brief Title: A Healthy Volunteer Study With Inhaled GSK573719 and Placebo
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 110106
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Healthy volunteers; New formulation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Active (Experimental): 100mcg 719
  Interventions: Drug: 100mcg
- Active 2 (Experimental): 500mcg '719
  Interventions: Drug: 500mcg
- Active 3 (Experimental): 1000mcg '719
  Interventions: Drug: 1000mcg
- Placebo (Placebo Comparator): Placebo '719
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 100mcg — 100mcg '719
  Arms: Active
Drug: 500mcg — 500mcg '719
  Arms: Active 2
Drug: 1000mcg — 1000mcg '719
  Arms: Active 3
Drug: Placebo — Placebo '719
  Arms: Placebo

SUMMARY:
This study is to look at a new formulation of GSK573719 to see if it is safe and tolerated in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy.
* Male or female 18 to 65 years of age inclusive.
* Non-childbearing women or women of child bearing potential who agree to use contraception
* Subject has had their CYP2D6 genotype confirmed and can be included in either of the following parts:
* Part 1: may include extensive, intermediate and ultra-rapid metabolizers
* Part 2: includes only poor (no enzyme activity) metabolizers, with previously confirmed phenotype
* Body Mass Index within the range 18 - 30 kg/m2 (inclusive).
* Capable of giving written informed consent
* Normal ECG;
* Normal lung function.
* Non-smokers (never smoked or not smoking for >6 months with <10 pack years history (Pack years = (cigarettes per day smoked/20) x number of years smoked))
* A signed and dated written informed consent is obtained from the subject
* The subject is capable of giving informed consent
* Available to complete the study

Exclusion Criteria:

* Any clinically important abnormality identified at the screening medical assessment (physical examination/medical history), clinical laboratory tests, or ECG (12-lead). 24hr Holter monitoring outside normal limits.
* A history of breathing problems (i.e. history of asthmatic symptomatology).
* Abnormal ECG.
* Abnormal blood pressure.
* Abnormal heart rate
* The subject has a positive pre-study drug/alcohol screen.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within three months of screening.
* A positive test for HIV antibody (if determined by the local SOPs).
* History of high alcohol consumption within three months of the study
* The subject has participated in a clinical trial and has received an IP within the following time period prior to the first dosing day in the current study: 30 days, five half-lives or twice the duration of the biological effect of the IP (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, (except for simple analgesics e.g. paracetamol), including vitamins, herbal and dietary supplements (including St John's Wort) within seven days (or 14 days if the drug is a potential enzyme inducer) or five half-lives (whichever is longer) prior to the first dose of study medication
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500mL within a 56 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Urinary cotinine levels indicative of smoking or history of regular use of tobacco- or nicotine-containing products prior to screening.
* The subject is unable to use the novel dry powder inhaler correctly.
* The subject has a known allergy or hypersensitivity to milk protein or the excipients magnesium stearate and lactose monohydrate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-05-05 (Actual); Primary Completion 2008-10-16 (Actual); Study Completion 2008-10-16 (Actual)

PRIMARY OUTCOMES:
General safety and tolerability endpoints: Adverse Events (AE), HR, BP, 12- lead ECG and lung function (FEV1) and clinical laboratory safety tests | Various

SECONDARY OUTCOMES:
Blood and urine levels of study drug | various

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Cahn A, Mehta R, Preece A, Blowers J, Donald A. Safety, tolerability and pharmacokinetics and pharmacodynamics of inhaled once-daily umeclidinium in healthy adults deficient in CYP2D6 activity: a double-blind, randomized clinical trial. Clin Drug Investig. 2013 Sep;33(9):653-64. doi: 10.1007/s40261-013-0109-6. PMID 23881566
- See also: Results for study 110106 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/110106?search=study&search_terms=110106#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 110106 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 110106 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 110106 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 110106 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 110106 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 110106 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 110106 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register